CLINICAL TRIAL: NCT05860595
Title: Evaluation the Safety and Efficacy of KL003 Cell Injection in the Treatment of Transfusion-dependent β-thalassemia.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: R&D Kanglin Biotech (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023021
Record Dates: First submitted 2023-05-08; First posted 2023-05-16 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-03

CONDITIONS: Transfusion-dependent Beta-Thalassemia
Keywords: Beta-Thalassaemia; Hematopoietic Stem-Cell Transplantation
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- KL003 cell injection Drug Product (Experimental): Each recruited subject will accept KL003 Transplantation.
  Interventions: Genetic: KL003 cell injection Drug Product

INTERVENTIONS:
Genetic: KL003 cell injection Drug Product — Transplant of auto-HSC transduced with lentiviral vector encoding βA-T87Q-globin gene.

SUMMARY:
This is a non-randomized, open-label, single-dose study. The aim of this study is to evaluate the safety and efficacy of the treatment with lentiviral vector encoding βA-T87Q-globin gene transduced autologous hematopoietic stem cells in subjects with transfusion-dependent β-thalassemia.

DETAILED DESCRIPTION:
Subject participation for this study will be 24 months. Subjects who enroll in this study will be asked to participate in a subsequent 13-year follow-up for gene therapy products.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age between 3-35 years
* Diagnosis of transfusion-dependent β-thalassemia and a history of at least 100 mL/kg/year of pRBCs or ≥8 transfusions of pRBCs per year for the prior 2 years
* Documented baseline, or pretransfusion, Hb level≤7 g/dL
* Karnofsky performance status ≥70 for subjects≥16 years of age; Lansky performance status of ≥70 for subjects<16 years of age
* Eligible to undergo auto-HSCT
* Willing and able to follow the research procedures and conditions, with good compliance
* Willing to receive at least the 2 years follow-up and maintain detailed medical records, including transfusion history
* Subject and/or legal guardians voluntarily participated in this clinical trial and signed the informed consent form, and can complete all follow-up in accordance with the protocol requirements

Exclusion Criteria:

* Subjects positive with the following etiological tests: human immunodeficiency virus(HIV-1-2), human cytomegalovirus (HCMV-DNA), EB virus (EBV-DNA), HBV (HBsAg/HBV-DNA positive), HCV antibody (HCV-Ab), Treponema pallidum antibody (TP-Ab)
* Clinically significant and active bacterial, viral, fungal, or parasitic infection as determined by the clinical investigator
* Contraindication to bone marrow collection
* Any prior or current malignancy or myeloproliferative or significant immunodeficiency disorder
* A white blood cell (WBC) count <3×10^9/L, and/or platelet count <100×10^9/L not related to hypersplenism
* Diagnosis of composite α thalassemia
* Participants with severe iron overload at the time of screening: severe iron overload of the liver showed by MRI, serum ferritin ≥ 5000 ng/mL, or moderate to severe iron overload of the heart
* Presence of unusual antibody of red blood cell antigens or tested positive for platelet antibody
* Meet the criteria for allo-HSCT and with an identified willing donor with a full HLA match
* Prior receipt of gene therapy or allo-HSCT
* Immediate family member (i.e. parent or siblings) with a known Familial Cancer Syndrome (including but not limited to hereditary breast and ovarian cancer syndrome, hereditary non-polyposis colorectal cancer syndrome and familial adenomatous polyposis)
* Diagnosis of a significant psychiatric disorder of the subject that could seriously impede the ability to participate in the study
* History of major organ damage including:

  1. Liver function test suggest AST or ALT levels >3× upper limit of normal (ULN);
  2. Total serum bilirubin value >2.5×ULN;if combined with Gilbert syndrome, total bilirubin >3×ULN and direct bilirubin value >2.5×ULN;
  3. History of bridging fibrosis, cirrhosis;
  4. Left ventricular ejection fraction <45%;
  5. New York Heart Association (NYHA) class III or IV congestive heart failure;
  6. Severe arrhythmia requiring medical treatment;
  7. Uncontrolled hypertension or unstable angina pectoris;
  8. Myocardial infarction or bypass or stent surgery within 12 months before drug administration;
  9. Valvular disease with clinical significance;
  10. Baseline calculated eGFR<60mL/min/1.73m2;
  11. Pulmonary function: FEV1/FVC<60% and/or diffusion capacity of carbon monoxide (DLco) <60% of prediction;
  12. Evidence of clinically significant pulmonary hypertension requiring medical intervention.
* Uncorrectable coagulation dysfunction or history of severe bleeding disorder
* Any other condition that would render the subject ineligible for HSCT, as determined by the attending transplant physician
* Known allergy to clinical trial drug (plerixafor or G-CSF or busulfan) or ingredient(DMSO etc.)
* Participation in another clinical study with an investigational drug within 30 days of Screening or participating in another clinical study with an investigational drug
* Inoculated live vaccine within 6 weeks prior to screening
* Pregnancy or breastfeeding women; Subjects or their sexual partners were unable to take medically recognized effective contraceptive measures during the 27-month study period
* The subjects or their parents would not comply with the study procedures outlined in the protocol
* Receipt of hydroxyurea therapy within 3 months before HSCT harvest
* Patients considered to be ineligible for the study by the investigator for reasons other than the above

Ages: 3 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2025-08-20 (Estimated); Study Completion 2025-10-24 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with successful lentiviral vector transduced CD34+ stem cell engraftment | Up to 42 days post transplant
  Successful engraftment was defined as neutrophil count [ANC] ≥0.5×10^9/L for 3 consecutive days
Engraftment time of neutrophil | Up to 42 days post transplant
  The first day when neutrophils ≥ 0.5×10^9/L for 3 consecutive days
Engraftment time of platelet | Up to 42 days post transplant
  The first day of platelet count ≥ 20.0×10^9/L for 7 consecutive days after platelet transfusion independence
Transplant-related mortality within 100 days and within 1 year after reinfusion of KL003 drug product | Up to 1 year post transplant
The number, frequency and severity of adverse events (AE) within 1 year after reinfusion of KL003 drug products | Up to 24 months post transplant
  Frequency and severity of AEs & SAEs identified according to NCI CTCAE 5.0

SECONDARY OUTCOMES:
The proportion of participants who meet the definition of transfusion independence (TI) for at least 6 months | Up to 24 months post transplant
  TI is defined as Hb ≥ 90.0 g/L after reinfusion and without disease-related routine blood transfusion for 6 months
The duration of transfusion independence | Up to 24 months post transplant
Changes in the frequency and volume of blood transfusion | Up to 24 months post transplant

CONTACTS AND LOCATIONS:
Locations (1):
- Regenerative Medicine Center, Tianjin, Tianjin Municipality, China